CLINICAL TRIAL: NCT00924937
Title: Randomized Clinical Trial on the Effects of Mediterranean Diet (Rich on Olive Oil) in the Reduction of Coronary Events of Patients With Coronary Disease
Brief Title: CORonary Diet Intervention With Olive Oil and Cardiovascular PREVention
Acronym: CORDIOPREV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitario Reina Sofia de Cordoba (Other Government)
Responsible Party: Principal Investigator, Francisco Perez Jimenez, Chief of Internal Medicine Unit, Hospital Universitario Reina Sofia de Cordoba
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CORDIOPREV
Record Dates: First submitted 2009-06-18; First posted 2009-06-19 (Estimated); Last update posted 2021-06-03 (Actual); Status verified 2021-05

CONDITIONS: Myocardial Infarction; Unstable Angina; Malignancy; Cognitive Decline; Diabetes Mellitus; Metabolic Syndrome
Keywords: Cardiovascular events; Blood pressure; Incidence of Cancer; Cognitive decline; Mediterranean Diet; Secondary Prevention; Low fat diet
MeSH Terms: conditions — Myocardial Infarction; Angina, Unstable; Neoplasms; Cognitive Dysfunction; Diabetes Mellitus; Metabolic Syndrome | interventions — Diet, Mediterranean; Diet, Fat-Restricted

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low Fat Diet (Active Comparator): Dietary Intervention with a Low fat diet: <30% fat (12% monounsaturated fatty acids; 6-8%polyunsaturated fatty acids; <10% saturated fatty acids)
  Interventions: Behavioral: Low Fat Diet
- Mediterranean Diet (Experimental): Dietary Intervention with a Mediterranean Diet: 35-38% fat (22% monounsaturated fatty acids; 6% polyunsaturated fatty acids; <10% saturated fatty acids).
  Interventions: Behavioral: Mediterranean Diet

INTERVENTIONS:
Behavioral: Mediterranean Diet — Mediterranean Diet:35-38% fat (22% MUFA; 6% PUFA; <10% SAT).
  Arms: Mediterranean Diet
Behavioral: Low Fat Diet — Low fat diet: <30% fat (12% MUFA; 6-8%PUFA; <10% SAT)
  Arms: Low Fat Diet

SUMMARY:
The purpose of this study is to compare the effects of the consumption of two different dietary patterns (low fat versus Mediterranean Diet) on the incidence of cardiovascular events of persons with coronary disease.

DETAILED DESCRIPTION:
Randomized clinical trial involving 1002 patients with coronary disease that are undergoing one of two diets in a randomized design (two groups; Mediterranean Diet 502 patients, Low Fat 500 patients) for 7 years. The two diets are: a)Low fat diet: <30% fat (12-14% monounsaturated fatty acids (MUFA); 6-8% polyunsaturated fatty acid (PUFA) ; <10% SAT) and b) Mediterranean Diet: >35% fat (22% MUFA; 6% PUFA ; <10% SAT).

Primary Objective:

Combined apparition of hard cardiovascular events (myocardial infarction, revascularization, ischemic stroke, documented peripheral artery disease or cardiovascular death).

Secondary Objectives:

Those related in the Outcome Measures section of this webpage

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent
* Clinical: Unstable coronary disease with documented vessel/myocardial damage

  * Acute Myocardial Infarction
  * Revascularization

Exclusion Criteria:

* Age < 20 or > 75 years (or life expectancy lower than 5 years).
* Patients already planned for revascularization.
* Patients submitted to revascularization in the last 6 months
* Grade II-IV Heart failure.
* Left ventricle dysfunction with ejection fraction lower than 35%.
* Patients unable to follow a protocol.
* Patients with severe uncontrol of Diabetes Mellitus, or those with Renal Insufficiency with plasma creatinine higher than 2mg/dl, or cerebral complications of Diabetes mellitus.
* Other chronic diseases:

  * Psychiatric diseases
  * Renal Insufficiency
  * Chronic Hepatopathy
  * Active Malignancy
  * Chronic obstructive pulmonary disease
  * Diseases of the digestive tract Endocrine disorders
* Patients participating in other Clinical trials (in the enrollment moment or 30 days prior).

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1002 (Actual)
Dates: Start 2009-11 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2021-05 (Actual)

PRIMARY OUTCOMES:
Combined apparition of hard cardiovascular events (myocardial infarction, revascularization, ischemic stroke, documented peripheral artery disease or cardiovascular death) after a median follow-up of 7 years. | Seven Years
  Combined apparition of hard cardiovascular events (myocardial infarction, revascularization, ischemic stroke, documented peripheral artery disease or cardiovascular death) after a median follow-up of 7 years.

SECONDARY OUTCOMES:
Evolution of arteriosclerosis: Evaluation of arteriosclerosis at different vascular beds. Silent arteriosclerosis. | Seven Years
  Data from clinical and/or diagnostic tests will be analyzed
Concentration of LDL cholesterol. | Seven Years
  Concentration of LDL cholesterol in blood samples
Atherogenic ratio, and Total cholesterol/HDL and LDL/HDL. | Seven Years
  Comparison of Atherogenic ratio, and Total cholesterol/HDL and LDL/HDL during the study
Metabolic control of carbohydrates (assessed by glycemic and insulin responses to intravenous tolerance test to glucose, basal glycemia and hba1c). | Seven Years
  Study of the metabolism of carbohydrates during the trial
Blood pressure. | Seven Years
  Study of blood pressure in response to the study
Incidence of malignancy. | Seven Years
  Appearance of malignancy
Progression of Cognitive Decline. | Seven Years
  Cognitive decline will be evaluated by validated questionnaires
Extended composite of cardiovascular disease progression | Seven Years
  Incidence of cardiac death, myocardial infarction, angina event, coronary revascularization or cardiac transplant, stroke, symptomatic heart failure, or any other clinical manifestation of cardiovascular event.
Extended composite of heart events | Seven Years
  Incidence of cardiac death , myocardial infarction , unstable angina , revascularization, heart failure, heart transplantation, cardiac arrest
Incidence of type 2 Diabetes Mellitus | Up to Seven Years
  Incidence of type 2 Diabetes Mellitus during the study
Anthropometric changes. Metabolic disease | Up to Seven Years
  Clinical features of metabolic disease: Metabolic Syndrome, Metabolic Phenotypes of Obesity or other classifications based on anthropometric features will be assessed during the study
Gut Microbiota | Up to Seven Years
  Changes in the percentage of different families of Microbiota will be analyzed during the study, and their impact on clinical events.
Arrhythmias | Up to Seven Years
  Study of relationship between existing or new Arrhythmias on clinical events
Individual evaluation of all components of the primary outcome. | Up to Seven Years
  Individual apparition of hard cardiovascular events:
  * myocardial infarction
  * revascularization
  * ischemic stroke
  * documented peripheral artery disease
  * cardiovascular death
Global Metabolomics | Up to Seven Years
  Global metabolomics in plasma, as well as techniques targeting specific sets of metabolites such as lipid-based lipid species, protein by proteomics, etc.
Specific metabolomics | Up to Seven Years
  Specific metabolomics in plasma fractions, specific bioparticles such as lipoproteins or specific cells, lipidomics, proteomics, targeted metabolomics, etc
Gene Expression | Up to Seven Years
  Changes in Gene Expression using transcriptomic techniques such as gene expression microarrays, quantitative PCR, GeneChip, etc
Inflammation and oxidative stress | Up to Seven Years
  Different physiological processes or metabolic pathways related to inflammation and oxidative stress will be studied
AGEs | Up to Seven Years
  Metabolism of advanced glycation end products.
Mineral metabolism | Up to Seven Years
  Impact of mineral metabolism on atherosclerosis
Echographic markers of cardiac function and clinical outcomes | Up to Seven Years
  Cardiac function studies by Echocardiography at baseline and during the study
Microparticles | Up to Seven Years
  Study of endothelial microparticles (vesicles formed from endothelial cells membrane after injury). The quantification of the EPCs and EMPs will be performed by flow cytometry
Subgroup analysis | Up to Seven Years
  27. Differential impact on certain subgroups: Sex, age, anthropometry, genetics, genomics, metabolism of immediate principles, cardiovascular risk factors, cancer, vascular function

OTHER OUTCOMES:
Endothelial function (Flow mediated dilation) | Up to Seven Years
  Endothelium response to ischemia in the brachial artery. Area under the curve, flow peak and time to maximum flow will be performed
genetics, genomics and epigenetics | Up to seven years
  Influence of genetic data in the development clinical outcomes
postprandial lipaemia | Up to seven years
  Postprandial lipemia study based on oral fat tolerance test depending on clinical and genetic variables
Study of other Clinical events | Up to seven years
  Clinical events not qualifying as primary endpoint nor in the secondary objectives 1 and 2, especially those associated with cardiovascular disease
Subgroup Studies | Up to seven years
  Differential impact on certain subgroups: Sex, age, anthropometry, genetics, genomics, metabolism of immediate principles, cardiovascular risk factors, cancer, vascular function
Further Studies | Up to Seven Years
  Additional secondary objectives will be carried out in light of current and/or future knowledge of ischemic heart disease risk factors, prognostic factors and pathophysiological pathways, and will include, but not be limited to, endothelial function, inflammation, cell biology, molecular biology, proteomics, genetics and epigenetics

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Perez-Jimenez, MD,PhD, Principal Investigator — Reina Sofia University Hospital
Locations (1):
- Reina Sofia University Hospital, Córdoba, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Delgado-Lista J, Alcala-Diaz JF, Torres-Pena JD, Quintana-Navarro GM, Arenas Larriva AP, Fuentes F, Garcia-Rios A, Yubero-Serrano EM, Rangel-Zuniga OA, Camargo A, Rodriguez-Cantalejo F, Katsiki N, Perez-Martinez P, Lopez-Miranda J; CORDIOPREV Investigators. Incidence of major adverse cardiovascular events decreases with greater adherence to both Mediterranean and low-fat dietary patterns in secondary prevention patients: a randomized controlled trial. Eur J Intern Med. 2026 Jan 28:106733. doi: 10.1016/j.ejim.2026.106733. Online ahead of print. PMID 41611577
- [Derived] Garcia-Rios A, Romero-Cabrera JL, Alcala-Diaz JF, Quintana-Navarro GM, Martin-Piedra L, Arenas-de Larriva AP, Torres-Pena JD, Rodriguez-Cantalejo F, Kales SN, Ordovas JM, Perez-Martinez P, Delgado-Lista J, Lopez-Miranda J. Long sleep duration pattern is associated with increased cardiovascular recurrence: Effect of long-term Mediterranean diet from the CORDIOPREV study. J Intern Med. 2025 Sep;298(3):237-250. doi: 10.1111/joim.20119. Epub 2025 Jul 17. PMID 40677148
- [Derived] Boughanem H, Gutierrez-Mariscal FM, Arenas-de Larriva AP, Torres-Pena JD, Romero-Cabrera JL, Rangel-Zuniga OA, Garcia-Fernandez H, Podadera-Herreros A, Rodriguez-Cantalejo F, Soehnlein O, Macias-Gonzalez M, Tinahones FJ, Yubero Serrano EM, Perez-Martinez P, Delgado-Lista J, Lopez-Miranda J. Effect of long-term Mediterranean versus low-fat diet on neutrophil count, and type 2 diabetes mellitus remission in patients with coronary heart disease: results from the CORDIOPREV study. Nutr Diabetes. 2025 Mar 27;15(1):11. doi: 10.1038/s41387-025-00360-3. PMID 40148287
- [Derived] Gutierrez-Mariscal FM, Lopez-Moreno A, Torres-Pena JD, Gomez-Luna P, Arenas-de Larriva AP, Romero-Cabrera JL, Luque RM, Uribarri J, Perez-Martinez P, Delgado-Lista J, Yubero-Serrano EM, Lopez-Miranda J. Modulation of circulating levels of advanced glycation end products and its impact on intima-media thickness of both common carotid arteries: CORDIOPREV randomised controlled trial. Cardiovasc Diabetol. 2024 Oct 14;23(1):361. doi: 10.1186/s12933-024-02451-4. PMID 39402581
- [Derived] Podadera-Herreros A, Arenas-de Larriva AP, Gutierrez-Mariscal FM, Alcala-Diaz JF, Ojeda-Rodriguez A, Rodriguez-Cantalejo F, Cardelo MP, Rodriguez-Cano D, Torres-Pena JD, Luque RM, Ordovas JM, Perez-Martinez P, Delgado-Lista J, Lopez-Miranda J, Yubero-Serrano EM. Mediterranean diet as a strategy for preserving kidney function in patients with coronary heart disease with type 2 diabetes and obesity: a secondary analysis of CORDIOPREV randomized controlled trial. Nutr Diabetes. 2024 May 16;14(1):27. doi: 10.1038/s41387-024-00285-3. PMID 38755195
- [Derived] Ojeda-Rodriguez A, Rangel-Zuniga OA, Arenas-de Larriva AP, Gutierrez-Mariscal FM, Torres-Pena JD, Romero-Cabrera JL, Podadera-Herreros A, Garcia-Fernandez H, Porras-Perez E, Luque RM, Kales SN, Perez-Martinez P, Delgado-Lista J, Yubero-Serrano EM, Lopez-Miranda J. Telomere length as biomarker of nutritional therapy for prevention of type 2 diabetes mellitus development in patients with coronary heart disease: CORDIOPREV randomised controlled trial. Cardiovasc Diabetol. 2024 Mar 16;23(1):98. doi: 10.1186/s12933-024-02175-5. PMID 38493287
- [Derived] Garcia-Fernandez H, Arenas-de Larriva AP, Lopez-Moreno J, Gutierrez-Mariscal FM, Romero-Cabrera JL, Molina-Abril H, Torres-Pena JD, Rodriguez-Cano D, Malagon MM, Ordovas JM, Delgado-Lista J, Perez-Martinez P, Lopez-Miranda J, Camargo A. Sex-specific differences in intestinal microbiota associated with cardiovascular diseases. Biol Sex Differ. 2024 Jan 19;15(1):7. doi: 10.1186/s13293-024-00582-7. PMID 38243297
- [Derived] Rivas-Garcia L, Quintana-Navarro GM, Torres-Pena JD, Arenas-de Larriva AP, Alcala-Diaz JF, Yubero-Serrano EM, Perez Caballero AI, Ortiz-Morales AM, Rangel-Zuniga OA, Lopez-Moreno A, Ordovas JM, Perez-Martinez P, Lopez-Miranda J, Delgado-Lista J. Dietary antioxidant intake reduces carotid intima-media thickness in coronary heart disease patients: From the CORDIOPREV study. Free Radic Biol Med. 2024 Jan;210:221-229. doi: 10.1016/j.freeradbiomed.2023.11.026. Epub 2023 Nov 29. PMID 38036071
- [Derived] Villasanta-Gonzalez A, Mora-Ortiz M, Alcala-Diaz JF, Rivas-Garcia L, Torres-Pena JD, Lopez-Bascon A, Calderon-Santiago M, Arenas-Larriva AP, Priego-Capote F, Malagon MM, Eichelmann F, Perez-Martinez P, Delgado-Lista J, Schulze MB, Camargo A, Lopez-Miranda J. Plasma lipidic fingerprint associated with type 2 diabetes in patients with coronary heart disease: CORDIOPREV study. Cardiovasc Diabetol. 2023 Aug 3;22(1):199. doi: 10.1186/s12933-023-01933-1. PMID 37537576
- [Derived] Gutierrez-Mariscal FM, Alcala-Diaz JF, Quintana-Navarro GM, de la Cruz-Ares S, Torres-Pena JD, Cardelo MP, Arenas-Larriva AP, Malagon MM, Romero-Cabrera JL, Ordovas JM, Perez-Martinez P, Delgado-Lista J, Yubero-Serrano EM, Lopez-Miranda J. Changes in quantity plant-based protein intake on type 2 diabetes remission in coronary heart disease patients: from the CORDIOPREV study. Eur J Nutr. 2023 Jun;62(4):1903-1913. doi: 10.1007/s00394-022-03080-x. Epub 2023 Mar 4. PMID 36869909
- [Derived] Mora-Ortiz M, Alcala-Diaz JF, Rangel-Zuniga OA, Arenas-de Larriva AP, Abollo-Jimenez F, Luque-Cordoba D, Priego-Capote F, Malagon MM, Delgado-Lista J, Ordovas JM, Perez-Martinez P, Camargo A, Lopez-Miranda J. Metabolomics analysis of type 2 diabetes remission identifies 12 metabolites with predictive capacity: a CORDIOPREV clinical trial study. BMC Med. 2022 Oct 27;20(1):373. doi: 10.1186/s12916-022-02566-z. PMID 36289459
- [Derived] Yubero-Serrano EM, Gutierrez-Mariscal FM, Gomez-Luna P, Alcala-Diaz JF, Perez-Martinez P, Lopez-Miranda J. Dietary modulation of advanced glycation end products metabolism on carotid intima-media thickness in type 2 diabetes patients: From the CORDIOPREV study. Clin Investig Arterioscler. 2023 May-Jun;35(3):105-114. doi: 10.1016/j.arteri.2022.08.004. Epub 2022 Sep 29. English, Spanish. PMID 36184301
- [Derived] Delgado-Lista J, Alcala-Diaz JF, Torres-Pena JD, Quintana-Navarro GM, Fuentes F, Garcia-Rios A, Ortiz-Morales AM, Gonzalez-Requero AI, Perez-Caballero AI, Yubero-Serrano EM, Rangel-Zuniga OA, Camargo A, Rodriguez-Cantalejo F, Lopez-Segura F, Badimon L, Ordovas JM, Perez-Jimenez F, Perez-Martinez P, Lopez-Miranda J; CORDIOPREV Investigators. Long-term secondary prevention of cardiovascular disease with a Mediterranean diet and a low-fat diet (CORDIOPREV): a randomised controlled trial. Lancet. 2022 May 14;399(10338):1876-1885. doi: 10.1016/S0140-6736(22)00122-2. Epub 2022 May 4. PMID 35525255
- [Derived] Cano-Ibanez N, Quintana-Navarro GM, Alcala-Diaz JF, Rangel-Zuniga OA, Camargo A, Yubero-Serrano EM, Perez-Corral I, Arenas-de Larriva AP, Garcia-Rios A, Perez-Martinez P, Delgado-Lista J, Lopez-Miranda J. Long-term effect of a dietary intervention with two-healthy dietary approaches on food intake and nutrient density in coronary patients: results from the CORDIOPREV trial. Eur J Nutr. 2022 Sep;61(6):3019-3036. doi: 10.1007/s00394-022-02854-7. Epub 2022 Mar 29. Erratum In: Eur J Nutr. 2022 Dec;61(8):4223-4225. doi: 10.1007/s00394-022-03006-7. PMID 35348875
- [Derived] Podadera-Herreros A, Alcala-Diaz JF, Gutierrez-Mariscal FM, Jimenez-Torres J, Cruz-Ares S, Arenas-de Larriva AP, Cardelo MP, Torres-Pena JD, Luque RM, Ordovas JM, Delgado-Lista J, Lopez-Miranda J, Yubero-Serrano EM. Long-term consumption of a mediterranean diet or a low-fat diet on kidney function in coronary heart disease patients: The CORDIOPREV randomized controlled trial. Clin Nutr. 2022 Feb;41(2):552-559. doi: 10.1016/j.clnu.2021.12.041. Epub 2022 Jan 6. PMID 35030530
- [Derived] Villasanta-Gonzalez A, Alcala-Diaz JF, Vals-Delgado C, Arenas AP, Cardelo MP, Romero-Cabrera JL, Rodriguez-Cantalejo F, Delgado-Lista J, Malagon MM, Perez-Martinez P, Schulze MB, Camargo A, Lopez-Miranda J. A plasma fatty acid profile associated to type 2 diabetes development: from the CORDIOPREV study. Eur J Nutr. 2022 Mar;61(2):843-857. doi: 10.1007/s00394-021-02676-z. Epub 2021 Oct 5. PMID 34609622
- [Derived] Jimenez-Torres J, Alcala-Diaz JF, Torres-Pena JD, Gutierrez-Mariscal FM, Leon-Acuna A, Gomez-Luna P, Fernandez-Gandara C, Quintana-Navarro GM, Fernandez-Garcia JC, Perez-Martinez P, Ordovas JM, Delgado-Lista J, Yubero-Serrano EM, Lopez-Miranda J. Mediterranean Diet Reduces Atherosclerosis Progression in Coronary Heart Disease: An Analysis of the CORDIOPREV Randomized Controlled Trial. Stroke. 2021 Nov;52(11):3440-3449. doi: 10.1161/STROKEAHA.120.033214. Epub 2021 Aug 10. Erratum In: Stroke. 2021 Nov;52(11):e754. doi: 10.1161/STR.0000000000000393. PMID 34372670
- [Derived] Vals-Delgado C, Alcala-Diaz JF, Roncero-Ramos I, Leon-Acuna A, Molina-Abril H, Gutierrez-Mariscal FM, Romero-Cabrera JL, de la Cruz-Ares S, van Ommen B, Castano JP, Ordovas JM, Perez-Martinez P, Delgado-Lista J, Camargo A, Lopez-Miranda J. A microbiota-based predictive model for type 2 diabetes remission induced by dietary intervention: From the CORDIOPREV study. Clin Transl Med. 2021 Apr;11(4):e326. doi: 10.1002/ctm2.326. No abstract available. PMID 33931973
- [Derived] Yubero-Serrano EM, Alcala-Diaz JF, Gutierrez-Mariscal FM, Arenas-de Larriva AP, Pena-Orihuela PJ, Blanco-Rojo R, Martinez-Botas J, Torres-Pena JD, Perez-Martinez P, Ordovas JM, Delgado-Lista J, Gomez-Coronado D, Lopez-Miranda J. Association between cholesterol efflux capacity and peripheral artery disease in coronary heart disease patients with and without type 2 diabetes: from the CORDIOPREV study. Cardiovasc Diabetol. 2021 Mar 25;20(1):72. doi: 10.1186/s12933-021-01260-3. PMID 33766036
- [Derived] Yubero-Serrano EM, Fernandez-Gandara C, Garcia-Rios A, Rangel-Zuniga OA, Gutierrez-Mariscal FM, Torres-Pena JD, Marin C, Lopez-Moreno J, Castano JP, Delgado-Lista J, Ordovas JM, Perez-Martinez P, Lopez-Miranda J. Mediterranean diet and endothelial function in patients with coronary heart disease: An analysis of the CORDIOPREV randomized controlled trial. PLoS Med. 2020 Sep 9;17(9):e1003282. doi: 10.1371/journal.pmed.1003282. eCollection 2020 Sep. PMID 32903262
- [Derived] Jimenez-Lucena R, Alcala-Diaz JF, Roncero-Ramos I, Lopez-Moreno J, Camargo A, Gomez-Delgado F, Quintana-Navarro GM, Vals-Delgado C, Rodriguez-Cantalejo F, Luque RM, Delgado-Lista J, Ordovas JM, Perez-Martinez P, Rangel-Zuniga OA, Lopez-Miranda J. MiRNAs profile as biomarkers of nutritional therapy for the prevention of type 2 diabetes mellitus: From the CORDIOPREV study. Clin Nutr. 2021 Mar;40(3):1028-1038. doi: 10.1016/j.clnu.2020.06.035. Epub 2020 Jul 15. PMID 32723508
- [Derived] Leon-Acuna A, Torres-Pena JD, Alcala-Diaz JF, Vals-Delgado C, Roncero-Ramos I, Yubero-Serrano E, Tinahones FJ, Castro-Clerico M, Delgado-Lista J, Ordovas JM, Lopez-Miranda J, Perez-Martinez P. Lifestyle factors modulate postprandial hypertriglyceridemia: From the CORDIOPREV study. Atherosclerosis. 2019 Nov;290:118-124. doi: 10.1016/j.atherosclerosis.2019.09.025. Epub 2019 Sep 28. PMID 31605877
- [Derived] Roncero-Ramos I, Alcala-Diaz JF, Rangel-Zuniga OA, Gomez-Delgado F, Jimenez-Lucena R, Garcia-Rios A, Vals-Delgado C, Romero-Baldonado C, Luque RM, Ordovas JM, Perez-Martinez P, Camargo A, Lopez-Miranda J. Prediabetes diagnosis criteria, type 2 diabetes risk and dietary modulation: The CORDIOPREV study. Clin Nutr. 2020 Feb;39(2):492-500. doi: 10.1016/j.clnu.2019.02.027. Epub 2019 Feb 21. PMID 30852029
- [Derived] Gomez-Marin B, Gomez-Delgado F, Lopez-Moreno J, Alcala-Diaz JF, Jimenez-Lucena R, Torres-Pena JD, Garcia-Rios A, Ortiz-Morales AM, Yubero-Serrano EM, Del Mar Malagon M, Lai CQ, Delgado-Lista J, Ordovas JM, Lopez-Miranda J, Perez-Martinez P. Long-term consumption of a Mediterranean diet improves postprandial lipemia in patients with type 2 diabetes: the Cordioprev randomized trial. Am J Clin Nutr. 2018 Nov 1;108(5):963-970. doi: 10.1093/ajcn/nqy144. PMID 30475968
- [Derived] Corina A, Rangel-Zuniga OA, Jimenez-Lucena R, Alcala-Diaz JF, Quintana-Navarro G, Yubero-Serrano EM, Lopez-Moreno J, Delgado-Lista J, Tinahones F, Ordovas JM, Lopez-Miranda J, Perez-Martinez P. Low Intake of Vitamin E Accelerates Cellular Aging in Patients With Established Cardiovascular Disease: The CORDIOPREV Study. J Gerontol A Biol Sci Med Sci. 2019 May 16;74(6):770-777. doi: 10.1093/gerona/gly195. PMID 30165472
- [Derived] Camargo A, Jimenez-Lucena R, Alcala-Diaz JF, Rangel-Zuniga OA, Garcia-Carpintero S, Lopez-Moreno J, Blanco-Rojo R, Delgado-Lista J, Perez-Martinez P, van Ommen B, Malagon MM, Ordovas JM, Perez-Jimenez F, Lopez-Miranda J. Postprandial endotoxemia may influence the development of type 2 diabetes mellitus: From the CORDIOPREV study. Clin Nutr. 2019 Apr;38(2):529-538. doi: 10.1016/j.clnu.2018.03.016. Epub 2018 Apr 11. PMID 29685478
- [Derived] Torres-Pena JD, Garcia-Rios A, Delgado-Casado N, Gomez-Luna P, Alcala-Diaz JF, Yubero-Serrano EM, Gomez-Delgado F, Leon-Acuna A, Lopez-Moreno J, Camargo A, Tinahones FJ, Delgado-Lista J, Ordovas JM, Perez-Martinez P, Lopez-Miranda J. Mediterranean diet improves endothelial function in patients with diabetes and prediabetes: A report from the CORDIOPREV study. Atherosclerosis. 2018 Feb;269:50-56. doi: 10.1016/j.atherosclerosis.2017.12.012. Epub 2017 Dec 8. PMID 29274507
- [Derived] Rangel-Zuniga OA, Cruz-Teno C, Haro C, Quintana-Navarro GM, Camara-Martos F, Perez-Martinez P, Garcia-Rios A, Garaulet M, Tena-Sempere M, Lopez-Miranda J, Perez-Jimenez F, Camargo A. Differential menopause- versus aging-induced changes in oxidative stress and circadian rhythm gene markers. Mech Ageing Dev. 2017 Jun;164:41-48. doi: 10.1016/j.mad.2017.04.002. Epub 2017 Apr 10. PMID 28408140
- [Derived] Gomez-Delgado F, Delgado-Lista J, Lopez-Moreno J, Rangel-Zuniga OA, Alcala-Diaz JF, Leon-Acuna A, Corina A, Yubero-Serrano E, Torres-Pena JD, Camargo A, Garcia-Rios A, Caballero J, Castano J, Ordovas JM, Lopez-Miranda J, Perez-Martinez P. Telomerase RNA Component Genetic Variants Interact With the Mediterranean Diet Modifying the Inflammatory Status and its Relationship With Aging: CORDIOPREV Study. J Gerontol A Biol Sci Med Sci. 2018 Mar 2;73(3):327-332. doi: 10.1093/gerona/glw194. PMID 27707805
- [Derived] Rangel-Zuniga OA, Corina A, Lucena-Porras B, Cruz-Teno C, Gomez-Delgado F, Jimenez-Lucena R, Alcala-Diaz JF, Haro-Mariscal C, Yubero-Serrano EM, Delgado-Lista J, Lopez-Moreno J, Rodriguez-Cantalejo F, Camargo A, Tinahones FJ, Ordovas JM, Lopez-Miranda J, Perez-Martinez P. TNFA gene variants related to the inflammatory status and its association with cellular aging: From the CORDIOPREV study. Exp Gerontol. 2016 Oct;83:56-62. doi: 10.1016/j.exger.2016.07.015. Epub 2016 Jul 29. PMID 27477483
- [Derived] Blanco-Rojo R, Delgado-Lista J, Lee YC, Lai CQ, Perez-Martinez P, Rangel-Zuniga O, Smith CE, Hidalgo B, Alcala-Diaz JF, Gomez-Delgado F, Parnell LD, Arnett DK, Tucker KL, Lopez-Miranda J, Ordovas JM. Interaction of an S100A9 gene variant with saturated fat and carbohydrates to modulate insulin resistance in 3 populations of different ancestries. Am J Clin Nutr. 2016 Aug;104(2):508-17. doi: 10.3945/ajcn.116.130898. Epub 2016 Jul 20. PMID 27440084
- [Derived] Leon-Acuna A, Alcala-Diaz JF, Delgado-Lista J, Torres-Pena JD, Lopez-Moreno J, Camargo A, Garcia-Rios A, Marin C, Gomez-Delgado F, Caballero J, Van-Ommen B, Malagon MM, Perez-Martinez P, Lopez-Miranda J. Hepatic insulin resistance both in prediabetic and diabetic patients determines postprandial lipoprotein metabolism: from the CORDIOPREV study. Cardiovasc Diabetol. 2016 Apr 19;15:68. doi: 10.1186/s12933-016-0380-y. PMID 27095446
- [Derived] Talavera-Garcia E, Delgado-Lista J, Garcia-Rios A, Delgado-Casado N, Gomez-Luna P, Gomez-Garduno A, Gomez-Delgado F, Alcala-Diaz JF, Yubero-Serrano E, Marin C, Perez-Caballero AI, Fuentes-Jimenez FJ, Camargo A, Rodriguez-Cantalejo F, Tinahones FJ, Ordovas JM, Perez-Jimenez F, Perez-Martinez P, Lopez-Miranda J. Influence of Obesity and Metabolic Disease on Carotid Atherosclerosis in Patients with Coronary Artery Disease (CordioPrev Study). PLoS One. 2016 Apr 11;11(4):e0153096. doi: 10.1371/journal.pone.0153096. eCollection 2016. PMID 27064675
- [Derived] Haro C, Montes-Borrego M, Rangel-Zuniga OA, Alcala-Diaz JF, Gomez-Delgado F, Perez-Martinez P, Delgado-Lista J, Quintana-Navarro GM, Tinahones FJ, Landa BB, Lopez-Miranda J, Camargo A, Perez-Jimenez F. Two Healthy Diets Modulate Gut Microbial Community Improving Insulin Sensitivity in a Human Obese Population. J Clin Endocrinol Metab. 2016 Jan;101(1):233-42. doi: 10.1210/jc.2015-3351. Epub 2015 Oct 27. PMID 26505825
- [Derived] Blanco-Rojo R, Alcala-Diaz JF, Wopereis S, Perez-Martinez P, Quintana-Navarro GM, Marin C, Ordovas JM, van Ommen B, Perez-Jimenez F, Delgado-Lista J, Lopez-Miranda J. The insulin resistance phenotype (muscle or liver) interacts with the type of diet to determine changes in disposition index after 2 years of intervention: the CORDIOPREV-DIAB randomised clinical trial. Diabetologia. 2016 Jan;59(1):67-76. doi: 10.1007/s00125-015-3776-4. Epub 2015 Oct 16. PMID 26474775
- [Derived] Perez-Martinez P, Alcala-Diaz JF, Delgado-Lista J, Garcia-Rios A, Gomez-Delgado F, Marin-Hinojosa C, Rodriguez-Cantalejo F, Delgado-Casado N, Perez-Caballero AI, Fuentes-Jimenez FJ, Camargo A, Tinahones FJ, Ordovas JM, Perez-Jimenez F, Lopez-Miranda J. Metabolic phenotypes of obesity influence triglyceride and inflammation homoeostasis. Eur J Clin Invest. 2014 Nov;44(11):1053-64. doi: 10.1111/eci.12339. PMID 25231836
- See also: Webpage of the study — http://www.cordioprev.es/index.php/en/